CLINICAL TRIAL: NCT01881750
Title: Pivotal Response Group Treatment for Parents of Young Children With Autism
Acronym: PRTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-11022010-7151
Record Dates: First submitted 2011-07-20; First posted 2013-06-20 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Autistic Disorder
Keywords: Autism PRT
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pivotal Response Training (PRT) (Experimental): 12 week program on instruction of Pivotal Response Training, consisting of group meetings and individual sessions.
  Interventions: Behavioral: Pivotal Response Training (PRT)
- Parent Education Group (PEG) (Placebo Comparator): 12 week program consisting of offering/discussion information for parents. No pivotal response training provided.
  Interventions: Behavioral: Parent Education Group (PEG)

INTERVENTIONS:
Behavioral: Pivotal Response Training (PRT) — 12 week program on instruction of Pivotal Response Training, consisting of group meetings and individual sessions.
  Arms: Pivotal Response Training (PRT)
Behavioral: Parent Education Group (PEG) — 12 week program consisting of offering/discussion information for parents. No pivotal response training provided.
  Arms: Parent Education Group (PEG)

SUMMARY:
This is a research study examining the effectiveness of pivotal response treatment group (PRTG) in targeting language skills in young children with autism. Research has demonstrated that behavioral interventions, such as Pivotal Response Training (PRT), lead to improvements in the core symptoms of autism. The purpose of this study is to further examine the effectiveness of teaching pivotal response treatment to parents of children with autism in a group format. To determine the effectiveness of pivotal response training group (PRTG) it will be compared to another parent education group by conducting a randomized controlled 12-week trial.

DETAILED DESCRIPTION:
This is a research study examining the effectiveness of pivotal response treatment group (PRTG) in targeting language skills in young children with autism. Research has demonstrated that behavioral interventions, such as Pivotal Response Training (PRT), lead to improvements in the core symptoms of autism. Researchers have begun to develop strategies to investigate the effectiveness of teaching parents how to implement PRT in a group format, as opposed to an individual format. Preliminary data has demonstrated that teaching PRT in a group format has shown to be effective in teaching parents and increasing children's communication skills. The purpose of this study is to further examine the effectiveness of teaching pivotal response treatment to parents of children with autism in a group format. To determine the effectiveness of pivotal response training group (PRTG) it will be compared to another parent education group by conducting a randomized controlled 12-week trial. PRTG will aim to teach parents pivotal response training strategies, whereas the parent psychoeducational group (PEG) will aim to teach parents information with regards to assessment and treatment for children with autism. By conducting this research it will improve researchers understanding of group treatment options for individuals with autism and allow us to help in the development of therapeutic approaches that can meet the increasing service demands for families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) based on Autism Diagnostic Interview - Revised (ADI-R), Autism Diagnostic Observation Schedule (ADOS), Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), and expert clinical opinion
* Outpatients between 2.0 and 6 years of age of either gender
* Children of all cognitive levels will be included as long as they are able to participate in the testing procedures to the extent that valid standard scores can be obtained
* Language delay as measured by the Preschool Language Scale 4th ed. (PLS-4)
* Participants must have the ability to make meaningful vocalizations, defined as the ability to make contingent vocalizations when prompted (i.e., vocal sound showing intent to communicate, but not necessarily clear words)
* Stable psychotropic medication(s) or biomedical interventions for at least one month prior to baseline measurements with no anticipated changes during study participation
* Stable behavioral treatment (Applied Behavioral Analysis, Floortime, or other interventions), speech therapy, and school placement for at least 2 months prior to baseline measurements with no expected changes during study participation
* No more than 60 minutes of 1:1 speech therapy per week
* The availability of at least one parent who can consistently participate in the group treatment and related activities of the research study
* Be male or female in good medical health
* Will be starting PRTG after the first magnetic resonance image (MRI) scan has occured and, if agreeable, blood draw or saliva sample
* Parents intend on continuing PRTG for a minimum of 12 weeks
* Parents must be 18 years of age or older.

Exclusion Criteria:

* A current or life-time diagnosis of severe psychiatric disorder (e.g., bipolar disorder…)
* A genetic abnormality, such as Fragile X, based on genetic testing, done as indicated
* Presence of active medical problem (e.g., unstable seizure disorder or heart disease)
* Participants taking psychotropic medications will not be included if their medications have not been stable for over a week
* Parents who do not have the ability to videotape parent and child interactions on a weekly basis
* Parents who are not willing to implement intervention strategies for at least one hour a day
* Parents who plan to alternate which parent attends the group sessions.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hardan AY, Gengoux GW, Berquist KL, Libove RA, Ardel CM, Phillips J, Frazier TW, Minjarez MB. A randomized controlled trial of Pivotal Response Treatment Group for parents of children with autism. J Child Psychol Psychiatry. 2015 Aug;56(8):884-92. doi: 10.1111/jcpp.12354. Epub 2014 Oct 27. PMID 25346345
- [Result] Gengoux GW, Berquist KL, Salzman E, Schapp S, Phillips JM, Frazier TW, Minjarez MB, Hardan AY. Pivotal Response Treatment Parent Training for Autism: Findings from a 3-Month Follow-Up Evaluation. J Autism Dev Disord. 2015 Sep;45(9):2889-98. doi: 10.1007/s10803-015-2452-3. PMID 25911977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred over 2 years (July 2010-June 2012). Participants were recruited through distribution of fliers at clinics and autism awareness events, referral by local professionals, and word of mouth.
Pre-assignment Details: One hundred and thirty-five potential subjects were screened after inquiring about the study; 104 signed a consent form. Forty one did not meet eligibility criteria and 10 decided not to participate before baseline measures.
Groups:
- Pivotal Response Training (PRT): Pivotal Response Training: 12 week program on instruction of Pivotal Response Training, consisting of group meetings and individual sessions.
- Parent Education Group (PEG): Parent Education Group: 12 week program consisting of offering/discussion information for parents. No pivotal response training provided.
Period: Overall Study
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Started | 27 | 26
Completed | 25 | 22
Not Completed | 2 | 4
Not completed — Changes in concomitant therapies | 2 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG) | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 26 | 53
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 21 | 20 | 41
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Communication During Structured Lab Observation (SLO) at 12 Weeks
Description: Total frequency of child's utterances during 10 minute videotaped SLO assessment.
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: Utterances
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 25 | 22
Utterances
  Baseline Total Utterances of SLO | 45.7 (23.1) | 40.8 (22.4)
  Week 12 Total Utterances of SLO | 64.5 (28.9) | 51.4 (33.8)
Statistical Analysis 1: Comparison: Pivotal Response Training (PRT) vs Parent Education Group (PEG); Group X Time Interaction Cohen's d; Test type: Superiority or Other; p = 0.42, Mixed Effects Regression Model

2. Secondary Outcome: Parenting Stress Index Total Score
Description: Higher Scores Mean higher stress level and lower scores mean less stress (Range: Minimum = 36; Maximum=180).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 92.04 (25.07) | 98.38 (26.97)
  12 Weeks | 90.91 (22.33) | 95.95 (28.53)

3. Secondary Outcome: Family Empowerment Scale Total Score
Description: Higher Scores Mean better/more empowered and lower scores mean worse/less empowered (Range: Minimum = 24; Maximum=170).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 127.78 (18.18) | 121.73 (19.91)
  Week 12 | 130.14 (18.78) | 121.68 (14.25)

4. Secondary Outcome: Behavior Rating Inventory of Executive Function- Preschool Global Executive Composite Score
Description: Higher scores indicate worse executive functioning and lower scores indicate better executive functioning (Range: Minimum=63; Maximum=189).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 124.19 (21.17) | 124.19 (24.69)
  Week 12 | 113.28 (21.44) | 119.91 (24.05)

5. Secondary Outcome: Repetitive Behavior Scale- Revised Total Score
Description: Higher total scores mean more repetitive behaviors and lower total scores mean fewer repetitive behaviors (Range: Minimum=0; Maximum=129).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 21.70 (14.62) | 26.23 (22.70)
  Week 12 | 20.04 (16.69) | 30.05 (24.78)

6. Secondary Outcome: Sensory Profile Questionnaire Sensory Seeking Raw Score
Description: Higher scores mean more typical sensory seeking behaviors and lower scores mean more abnormal sensory seeking behaviors (Range: Minimum=0; Maximum=85).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 25
score on a scale
  Baseline | 60.81 (9.51) | 60.92 (12.02)
  Week 12 | 61.52 (11.09) | 65.52 (11.86)

7. Secondary Outcome: Pediatric Quality of Life Scale Scaled Total Mean Score
Description: Higher scores mean better quality of life and lower scores mean worse quality of life (Range: Minimum=0; Maximum=100).
Time Frame: Baseline, 12 weeks
Population: Participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Number analyzed (Participants) | 27 | 26
score on a scale
  Baseline | 64.86 (15.72) | 67.18 (15.66)
  Week 12 | 67.38 (14.06) | 67.45 (16.26)

ADVERSE EVENTS:
Arm/Group | Pivotal Response Training (PRT) | Parent Education Group (PEG)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26

LIMITATIONS AND CAVEATS:
The moderate sample size meant that power to detect complex multicomponent patterns was limited. There is also no information available about longer term effects of the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No